CLINICAL TRIAL: NCT06925750
Title: An Open-label Extension Study to Evaluate Safety and Tolerability of Sotatercept (MK-7962) Administered Using a Weight-banded Approach in Participants With Pulmonary Arterial Hypertension (PAH) on Standard of Care
Brief Title: A Clinical Study of Sotatercept (MK-7962) in People With Pulmonary Arterial Hypertension (MK-7962-031/LIGHTRAY EXTENSION)
Acronym: LIGHTRAY EXT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7962-031; MK-7962-031 (Other: MSD); 2024-518687-12-00 (Registry Identifier: EU CT); U1111-1314-0614 (Registry Identifier: UTN); jRCT2061250021 (Registry Identifier: jRCT (Japan Registry of Clinical Trials))
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Weight-banded sotatercept dosing (Experimental): Participants will receive sotatercept via subcutaneous (SC) injection every 3 weeks at an initial dose of up to 45 mg and then at a maintenance dose of up to 90 mg using a weight-banded method and will continue treatment for up to 24 months. All eligible participants will receive weight-banded dosing at the dosing level (initial or maintenance) at which they finished MK-7962-024 (LIGHTRAY). Participants will continue to take their background PAH therapy during the study.
  Interventions: Biological: Sotatercept; Drug: Background PAH Therapy

INTERVENTIONS:
Biological: Sotatercept — SC injection administered every 3 weeks
  Other Names: MK-7962; ACE-011
Drug: Background PAH Therapy — Background PAH therapy may consist of the following drug classes: single, double, or triple combination of therapy with endothelin-receptor antagonists, phosphodiesterase inhibitors, soluble guanylate cyclase stimulators, and/or prostacyclin analogs or receptor antagonists

SUMMARY:
Researchers are looking for other ways to treat pulmonary arterial hypertension (PAH). Sotatercept is a study medicine that is designed to treat PAH.

A past study, MK-7962-024 (LIGHTRAY) (NCT06664801), learned about the safety and effects of sotatercept in people with PAH. One of the goals of that study was to learn about sotatercept when given at a dose (amount) based on the weight range a person is in (weight-banded doses) compared to when given based on a person's exact weight.

This is an extension study, which means people who took part in MK-7962-024 (LIGHTRAY) may be able to join this study. In this extension study, people will get weight-banded doses of sotatercept. The main goal of this study is to learn about the safety of weight-banded doses of sotatercept and if people tolerate it over a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has completed the treatment period of study MK-7962-024 (LIGHTRAY) (including Visit 11) on study intervention, did not discontinue study intervention, and is able to safely enroll into MK-7962-031 (LIGHTRAY EXTENSION)
* Has not started treatment with commercially available sotatercept

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

- Has current exposure or is planning to begin treatment with an activin signaling inhibitor (other than sotatercept)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-06-16 (Estimated); Study Completion 2028-06-16 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 28 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants who Discontinue Study Intervention Due to an AE | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study intervention due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (73):
- United States (3):
  - University of Colorado Anschutz Medical Campus-University of Colorado Hospital Cardiac and Vascular ( Site 1930), Aurora, Colorado
  - University of Kansas Medical Center ( Site 1928), Kansas City, Kansas
  - University of New Mexico Health Sciences Center - Department of Internal Medicine ( Site 1916), Albuquerque, New Mexico
- Argentina (5):
  - Centro Medico Capital ( Site 0002), La Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 0006), Mar del Plata, Buenos Aires
  - Instituto Medico Rio Cuarto ( Site 0010), Río Cuarto, Córdoba Province
  - Instituto de Cardiologia Juana F. Cabral ( Site 0008), Corrientes
  - Hospital Provincial Jose Maria Cullen ( Site 0005), Santa Fe
- Australia (4):
  - Royal Prince Alfred Hospital ( Site 0103), Camperdown, New South Wales
  - Westmead Hospital ( Site 0100), Westmead, New South Wales
  - Wesley Research Institute ( Site 0101), Auchenflower, Queensland
  - The Alfred Hospital ( Site 0102), Melbourne, Victoria
- IUCPQ ( Site 0208), Québec, Quebec, Canada
- China (4):
  - Guangdong Provincial People's Hospital-Cardiology ( Site 2000), Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University ( Site 2002), Changsha, Hunan
  - Shanghai Pulmonary Hospital ( Site 2004), Shanghai, Shanghai Municipality
  - Yan an Hospital of Kunming City ( Site 2011), Kunming, Yunnan
- Colombia (4):
  - Clinica Colsanitas - Sede Reina Sofia ( Site 0303), Bogotá, Bogota D.C.
  - Fundacion Santa Fe de Bogota ( Site 0302), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 0301), Montería, Departamento de Córdoba
  - Clínica Imbanaco S.A.S ( Site 0304), Cali, Valle del Cauca Department
- Vseobecna fakultni nemocnice v Praze ( Site 0400), Prague, Praha 2, Czechia
- France (4):
  - CHU Bordeaux Haut-Leveque ( Site 0501), Pessac, Aquitaine
  - C.H.U Hôpital Nord ( Site 0500), Marseille, Bouches-du-Rhone
  - CHU de Rouen ( Site 0503), Rouen, Haute-Normandie
  - CHU GABRIEL MONTPIED ( Site 0504), Clermont-Ferrand, Puy-de-Dome
- Hungary (3):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ-Családorvosi Intézet és Rendelő ( Site 0704), Szeged, Csongrád megye
  - Semmelweis Egyetem ( Site 0701), Budapest, Pest County
  - Gottsegen György Országos Kardiovaszkuláris Intézet ( Site 0702), Budapest, Pest County
- Israel (4):
  - Rambam Health Care Campus ( Site 0802), Haifa
  - Carmel Hospital ( Site 0803), Haifa
  - Rabin Medical Center ( Site 0805), Petah Tikva
  - Sheba Medical Center ( Site 0801), Ramat Gan
- Italy (7):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico ( Site 0902), Milan, Lombardy
  - Azienda Ospedaliera Universitaria Integrata ( Site 0908), Verona, Veneto
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 0905), Bologna
  - Ospedale San Martino ( Site 0901), Genova
  - Fondazione IRCCS Policlinico San Matteo ( Site 0909), Pavia
  - AOU Policlinico Umberto I ( Site 0910), Roma
  - Ospedale Civile SS Annunziata ( Site 0903), Sassari
- Japan (6):
  - Nagoya University Hospital ( Site 2102), Nagoya, Aichi-ken
  - National Cerebral and Cardiovascular Center ( Site 2103), Suita, Osaka
  - The University of Tokyo Hospital ( Site 2101), Bunkyo, Tokyo
  - Kyorin University Hospital ( Site 2100), Mitaka, Tokyo
  - Kyushu University Hospital ( Site 2105), Fukuoka
  - National Hospital Organization Okayama Medical Center ( Site 2104), Okayama
- Netherlands (2):
  - Radboud University Medical Center ( Site 1001), Nijmegen, Gelderland
  - Sint Antonius Ziekenhuis ( Site 1000), Nieuwegein, Utrecht
- Singapore (2):
  - National University Heart Centre, Singapore ( Site 1200), Singapore, Central Singapore
  - National Heart Centre Singapore ( Site 1201), Singapore, Central Singapore
- South Korea (6):
  - Chonnam National University Hospital ( Site 1304), Gwangju, Kwangju-Kwangyokshi
  - Pusan National University Hospital ( Site 1305), Seogu, Pusan-Kwangyokshi
  - Seoul National University Hospital ( Site 1302), Seoul
  - Severance Hospital Yonsei University Health System ( Site 1300), Seoul
  - Asan Medical Center ( Site 1303), Seoul
  - Samsung Medical Center ( Site 1301), Seoul
- Spain (8):
  - Hospital Universitari Son Espases ( Site 1412), Palma, Balearic Islands
  - Hospital Universitario Marqués de Valdecilla ( Site 1405), Santander, Cantabria
  - Hospital Clinic de Barcelona ( Site 1406), Barcelona, Catalonia
  - Hospital Universitari Vall d''Hebron ( Site 1404), Barcelona
  - Hospital Universitario 12 de Octubre ( Site 1403), Madrid
  - Hospital Universitario La Paz ( Site 1410), Madrid
  - Hospital Universitario Virgen del Rocio ( Site 1407), Seville
  - HOSPITAL GENERAL UNIVERSITARIO DE TOLEDO ( Site 1408), Toledo
- Taiwan (2):
  - National Cheng Kung University Hospital ( Site 1501), Tainan
  - Taipei Veterans General Hospital ( Site 1502), Taipei
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital ( Site 1600), Bangkoknoi, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital ( Site 1601), Muang, Chiang Mai
- United Kingdom (5):
  - Royal Papworth Hospital ( Site 1802), Cambridge, Cambridgeshire
  - Royal Free Hospital ( Site 1803), London, England
  - Royal Brompton Hospital ( Site 1804), London, London, City of
  - Hammersmith Hospital ( Site 1801), London, London, City of
  - Golden Jubilee National Hospital ( Site 1800), Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com